CLINICAL TRIAL: NCT06932263
Title: A Phase IIb, Multicentre, Double-blind, Placebo-controlled Dose Range Finding Study to Assess Efficacy and Safety of Tozorakimab in Adult Participants With Uncontrolled Asthma on Medium-to High Dose Inhaled Corticosteroids
Brief Title: Dose Range Finding Study to Assess Efficacy and Safety of Tozorakimab in Adults With Uncontrolled Asthma on Medium-to-High Dose Inhaled Corticosteroids
Acronym: Umbriel
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9181C00002; 2024-519116-14-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is a parallel-group treatment study with 3 arms. Participants will be randomised in a ratio of 1:1:1 to one of the 3 treatment arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tozorakimab Dose 1 (Experimental): Dosing subcutaneously tozorakimab Dose 1
  Interventions: Drug: Tozorakimab
- Tozorakimab Dose 2 (Experimental): Dosing subcutaneously tozorakimab Dose 2 and placebo
  Interventions: Drug: Tozorakimab
- Placebo (Placebo Comparator): Dosing subcutaneously with equivalent volume to tozorakimab
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tozorakimab — The drug will be administered subcutaneously.
  Arms: Tozorakimab Dose 1; Tozorakimab Dose 2
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Placebo

SUMMARY:
This is a dose-range finding, double-blind, placebo-controlled, phase IIb study designed to assess efficacy and safety of tozorakimab administered subcutaneously in adult participants with uncontrolled asthma receiving medium-to-high dose inhaled corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study-specific procedures.
2. Adults aged 18-75, inclusive when signing the informed consent.
3. Documented physician-diagnosis of asthma for at least 12 months.
4. Treated with medium or high dose ICS in combination with LABA.
5. Demonstration of uncontrolled asthma through ACQ-6 score ≥ 1.5 .
6. Pre-bronchodilator FEV1 ≥ 40% to ≤ 90% of predicted normal.
7. Documented exacerbation history in the last 12 months and biomarker requirements of:

   1. 2 severe exacerbations OR
   2. 1 severe exacerbation and:

   (i) Eosinophils ≥ 150 cells/µl or (ii) FeNo ≥ 25 ppb
8. Participants need to demonstrate a ≥70% compliance for Asthma Daily Diary.
9. Women of Child Bearing Potential (WOCBP) must have a negative pregnancy test.
10. Contraceptive use by males and females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Completed treatment for respiratory infection with antibiotics in the 4 weeks prior to Visit 1.
2. Clinically significant pulmonary disease other than asthma .
3. Current smokers, former smokers with >10 pack-years history.
4. Clinically significant aortic stenosis or pulmonary arterial hypertension.
5. Active tuberculosis, hepatitis, HIV, or current diagnosis of cancer or immune complex disease.
6. Unstable cardiovascular disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2027-06-24 (Estimated); Study Completion 2028-03-16 (Estimated)

PRIMARY OUTCOMES:
Annualised rate of severe asthma exacerbations | Over 26 to 52 weeks
  The rate ratio of severe asthma exacerbations will be assessed in the participants with uncontrolled moderate-to-severe asthma and ≥ 1 severe exacerbation within 12 months prior to screening.

SECONDARY OUTCOMES:
Annualised rate of severe asthma exacerbations | Over 26 to 52 weeks
  The rate ratio of severe asthma exacerbations will be assessed in the participants with uncontrolled moderate-to-severe asthma and baseline eosinophils < 300 cells/µL and history of ≥2 severe exacerbations within 12 months prior to screening.
Time to first severe asthma exacerbation | Over 26 to 52 weeks
  To evaluate the effect of two dose levels of tozorakimab compared to placebo on time to first severe asthma exacerbations.
Change from baseline in pre-bronchodilator forced expiratory volume in 1 second (FEV1) | Over weeks 20 to 26
  Difference in mean change from baseline between tozorakimab and placebo.
Change from baseline in post-bronchodilator FEV1 | At week 26
  Difference in mean change from baseline between tozorakimab and placebo.
Change from baseline in the Asthma Control Questionnaire 6 (ACQ-6) | At week 26
  Difference in mean change from baseline between tozorakimab and placebo. The ACQ-6 has 6 questions (regarding asthma symptoms and rescue bronchodilator use). Answering the questions results in a score out of 6. A Score of 0 indicates complete control and 6 reflects severely uncontrolled disease.
Change from baseline in the Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ12+) | At week 26
  Difference in mean change from baseline between tozorakimab and placebo. The AQLQ12+ includes 32 questions grouped into four domains: symptoms; activity limitations; emotional function; and, environmental stimuli. Each question is scored on a seven-point Likert scale, which ranges from 7 (no impairment) to 1 (severe impairment). The overall score is calculated as the mean of all questions, and the four domain scores are the means of the scores for the questions in the respective domains.
Trough serum concentrations of tozorakimab | Over 52 weeks
  Pharmacokinetics: concentrations of tozorakimab in trough serum.
Anti-drug antibody incidence | Over 52 weeks
  Immunogenicity: Number of Participants With Positive Antibodies to tozorakimab

CONTACTS AND LOCATIONS:
Locations (176):
- United States (49):
  - Research Site, Bakersfield, California
  - Research Site, Huntington Beach, California
  - Research Site, La Mesa, California
  - Research Site, Newport Beach, California
  - Research Site, San Jose, California
  - Research Site, Wilmington, Delaware
  - Research Site, Cutler Bay, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palmetto Bay, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Boise, Idaho
  - Research Site, Indianapolis, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, White Marsh, Maryland
  - Research Site, Farmington Hills, Michigan
  - Research Site, Warren, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Grand Island, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Toms River, New Jersey
  - Research Site, Maspeth, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Kings Mountain, North Carolina
  - Research Site, Toledo, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Grants Pass, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, DuBois, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, Rock Hill, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Forney, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Tyler, Texas
  - Research Site, Victoria, Texas
  - Research Site, Roy, Utah
  - Research Site, Bellingham, Washington
  - Research Site, Kingwood, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (6):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, La Plata
  - Research Site, Mendoza
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
- Brazil (8):
  - Research Site, Caxias do Sul
  - Research Site, Criciúma
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Chile (5):
  - Research Site, Curicó
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (14):
  - Research Site, Baotou
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Huizhou
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Wenzhou
  - Research Site, Xuzhou
- France (7):
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Pessac
  - Research Site, Strasbourg
  - Research Site, Suresnes
- Greece (4):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (6):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gödöllő
  - Research Site, Pécs
  - Research Site, Törökbálint
- India (10):
  - Research Site, Belagavi
  - Research Site, Coimbatore
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Faridabad
  - Research Site, Gūrgaon
  - Research Site, Kochi
  - Research Site, Lucknow
  - Research Site, New Delhi
  - Research Site, Vadodara
- Israel (4):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
- Italy (4):
  - Research Site, Catania
  - Research Site, Foggia
  - Research Site, Genoa
  - Research Site, Roma
- Japan (14):
  - Research Site, Fukuoka
  - Research Site, Ginowan-shi
  - Research Site, Hiroshima
  - Research Site, Ishinomaki
  - Research Site, Kawaguchi-shi
  - Research Site, Kiyose-shi
  - Research Site, Kobe
  - Research Site, Meguro-ku
  - Research Site, Miura
  - Research Site, Neyagawa
  - Research Site, Sapporo
  - Research Site, Takamatsu
  - Research Site, Ube
  - Research Site, Yokohama
- Research Site, Lima, Peru
- Philippines (6):
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Lipa City
  - Research Site, Manadaluyong City
  - Research Site, Quezon City
  - Research Site, Roxas City
- South Africa (7):
  - Research Site, Benoni
  - Research Site, Brackenfell
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Somerset West
  - Research Site, Tygervalley
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Seoul
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Patraix
  - Research Site, Santander
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (6):
  - Research Site, Bangkok
  - Research Site, Chanthaburi
  - Research Site, Chiang Rai
  - Research Site, Chon Buri
  - Research Site, Khon Kaen
  - Research Site, Nakhon Sri Thammarat
- Turkey (Türkiye) (7):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Kayseri
  - Research Site, Mersin
- Vietnam (5):
  - Research Site, Da Nang
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/